CLINICAL TRIAL: NCT05908123
Title: The Blank Center CARE Model™: An Anti-Ableist Approach to Treatment
Brief Title: Exploring the Nature, Assessment and Treatment of Stuttering
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015050044
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stuttering; Stuttering, Adult; Stuttering, Childhood; Stuttering, Developmental
Keywords: stuttering, communication competence, adult, treatment
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blank Center CARE Model (Communication, Advocacy, Resilience, Education) (Experimental)
  Interventions: Behavioral: The Blank Center CARE Model(TM) for Individuals who Stutter

INTERVENTIONS:
Behavioral: The Blank Center CARE Model(TM) for Individuals who Stutter — The over-arching goal of the Blank Center CARE Model is to ensure individuals who stutter communicate effectively, advocate for themselves in a manner that maintains agency, and ensure their quality of life does not depend on producing, or attempting to control, stuttered speech.
  Other Names: Communication-Centered Treatment (CCT)

SUMMARY:
The purposes of this study are to 1) investigate potential speech, language, and psychosocial contributions to the experience of stuttering in monolingual and multilingual speakers, and to 2) evaluate interdisciplinary, telehealth, and speech-language pathology treatment methods and clinical training specific to fluency disorders.

DETAILED DESCRIPTION:
Stuttering is a neurophysiological communication disorder characterized by a disruption in the forward flow of speech. Stuttering is multifactorial in nature, meaning there are several factors that likely to contribute to the development of stuttering in children and persistence of stuttering into adulthood. About 1% of the worldwide population stutters. In the United States, over 3 million people stutter. Research suggests people who stutter present with negative cognitive and affective components of the disorder, and that the general population holds negative perceptions of stuttering. Historically, people who stutter spend thousands of dollars on treatment that is not effective in mitigating the negative impact of stuttering on their overall communication and quality of life.

Speech-language pathologists evaluate and treat persons who stutter across the lifespan. Research suggests speech-language pathologists report fluency disorders (stuttering and cluttering) as the communication disorders with which they feel least competent and comfortable.

Thus, the purposes of this study are to 1) investigate potential speech, language, psychosocial, and motor contributions to stuttered speech production in monolingual and multilingual speakers and to 2) evaluate interdisciplinary, telehealth, and speech-language pathology treatment methods and clinical training tools specific to fluency disorders.

ELIGIBILITY:
Inclusion Criteria:

A participant will be considered a child who stutters (ages 2-17 years) if

* their parent/caregiver reports concern that their child is a person who stutters,
* they exhibit three of more stuttering-like disfluencies (e.g., sound/syllable repetitions, (in)audible sound prolongations, whole-word repetitions) per 300-word speech sample, or
* they present with an overall score of 11 or higher on the Stuttering Severity Instrument - 4th Edition (SSI-4).

A participant will be considered an adult who stutters (18+ years) if

* they report they are a person who stutters,
* they have received a formal diagnosis of stuttering from a certified speech-language pathologist,
* they exhibit three of more stuttering-like disfluencies (e.g., sound/syllable repetitions, (in)audible sound prolongations, whole-word repetitions) per 300-word speech sample, or
* they present with an overall score of 11 or higher on the Stuttering Severity Instrument - 4th Edition (SSI-4).

Exclusion Criteria:

• There are no exclusion criteria for persons who stutter.

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2015-05-22 (Actual); Primary Completion 2035-05-22 (Estimated); Study Completion 2035-05-22 (Estimated)

PRIMARY OUTCOMES:
Communication Competence | 11-weeks
  psychometric measures of communication competence (e.g., CARE Assessment: Communication Subscale)
Advocacy | 11-weeks
  psychometric measures of self-advocacy (e.g., CARE Assessment: Advocacy Subscale)
Resilience | 11-weeks
  psychometric measures of resilience (e.g., CARE Assessment: Resilience Subscale)
Education | 11-weeks
  psychometric measures of education about stuttering (e.g., CARE Assessment: Education Subscale)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney T Byrd, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- Arthur M. Blank Center for Stuttering Education and Research, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: primary website for research center [Arthur M. Blank Center for Stuttering Education and Research] — https://blankcenterforstuttering.org/